CLINICAL TRIAL: NCT04960800
Title: Effect of a Specific Exercise Program During Pregnancy on Diastasis Recti Abdominis: Study Protocol for a Randomized Controlled Trial
Brief Title: Effect of a Specific Exercise Program During Pregnancy on Diastasis Recti Abdominis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bergen (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101944102
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Diastasis Recti Abdominis; Pregnancy Related
Keywords: pregnancy; ultrasonography; exercise; diastasis recti abdominis; inter-recti distance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This will be an exploratory, assessor blinded, randomized, controlled, parallel group trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: To ensure randomization to the two groups in the RCT, participants will, following baseline assessments, be allocated to the two groups by block randomization. Blocking will be masked and not stated in the protocol to avoid selection bias. The group allocation will be administrated by a research assistant, to ensure blinding of the assessor. This study is assessor blinded only, as participants and the physiotherapist running the intervention groups cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the intervention group will participate in a 12- week specific exercise programme led by an experienced women's health physiotherapist. These groups will take place at a private physiotherapy clinic twice a week. In addition, the participants will carry out a self-managed exercise program twice weekly for the same 12-week period. They will be provided with an exercise diary so that adherence to the intervention can be registered and monitored. This exercise diary will be sent to the participants once a week as an electronic questionnaire; this will ensure that the information recorded is standardized and that the research assistant can aid the participants to register their activity and encourage the participants to adhere to the intervention.
  Interventions: Other: Specific exercises
- Control group (No Intervention): The control group will not participate in any exercise intervention. The participants in the control group will be explained the importance of a control group in RCTs and will be recommended to continue with their normal activity levels. They will however, be recommended to follow national guidelines for general exercise during pregnancy and will receive information about these guidelines (15).

INTERVENTIONS:
Other: Specific exercises — Specific exercises which aims to contract the recti abdominis combined with functional exercises with the aim to contract all the layers of the anterior abdominal wall. Strengthening dosage will be applied with 3 sets, containing between 8 and 12 repetitions of maximal load.
  Arms: Intervention group

SUMMARY:
Diastasis Rectus abdominis is a common condition in pregnant and postpartum women, where the connective tissue between the two muscle bellies of the rectus abdominis muscle is stretched and weakened, causing an increased inter-rectus distance. Treatment of this condition aim to reduce the inter-rectus distance, and conservative treatment including therapeutic exercise is the primary treatment of choice. To date, there is no generally accepted protocol of therapeutic exercises for this condition, and the evidence as to which exercise modality is the most effective and feasible in reducing the inter-rectus distance in women presenting with diastasis rectus abdominis is both sparse and weak. As this condition occur during the last two trimesters of pregnancy and as there is a paucity of high-quality studies on a pregnant population, investigators will conduct a randomized controlled trial on the effect of a specific exercise program during pregnancy on diastasis rectus abdominis.

100 pregnant women in gestation week 25 presenting with diastasis rectus abdominis of ≥ 28 mm will be included. Participants will be allocated to either an intervention group or a control group by block randomization. The intervention group will participate in a 12-week specific exercise program, consisting of two group sessions and two self-managed sessions weekly. The control group will not participate in any exercise intervention; however, participants will be recommended to follow national guidelines for general exercise during pregnancy. Participants will be assessed prior to intervention, post intervention at gestation week 37, and 6 weeks, 6 and 12 months postpartum. The primary outcome measure will be change in the inter-rectus distance in mm, measured by two-dimensional ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* healthy pregnant women
* in gestation week 25
* presenting with an inter-rectus distance of 28 mm or more at the level of the umbilicus, and/or 2 cm above and below the umbilicus at rest on initial assessment. Participants presenting with a protrusion along the Linea Alba will also be included, even if they do not meet the inclusion criteria with an inter-rectus distance of 28 mm or more
* Both primi- and multigravida women will be included, and there will be no limitations on number of fetuses

Exclusion Criteria:

* pregnancies where exercise is contraindicated
* serious illnesses regarding both mother and fetus
* inability to understand Scandinavian languages
* failure to complete and present an informed consent form
* presence of chronic physical or mental illness incompatible with the intervention

Exclusion criteria during the study period is stillbirth or premature birth before gestation week 37; onset of serious illnesses regarding both mother and foetus; and pregnancies where exercise is contraindicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be change in inter-rectus distance in mm, measured by two-dimensional ultrasonography. | All participants will be assessed prior to intervention start in gestation week 27. They will then be reassessed at end of the intervention period at gestation week 37. Assessments will also be done 6 weeks, 6 and 12 months postpartum.
  The inter-rectus distance is the distance between the two muscle bulks of the rectus abdominis muscle. As the two muscle bulks are connected through the connective tissue Linea Alba, the inter-rectus distance is equivalent to the width of the line alba.The inter-rectus distance is measured 2 cm above and 2 cm below the umbilicus. Images of the inter-rectus distance is taken using 2-dimensional ultrasound, and measured using the free Microdicom software. Measurements will be done in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Haukenes, PhD, Study Director — University of Bergen
Locations (1):
- University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Theodorsen NM, Bo K, Fersum KV, Haukenes I, Moe-Nilssen R. Pregnant women may exercise both abdominal and pelvic floor muscles during pregnancy without increasing the diastasis recti abdominis: a randomised trial. J Physiother. 2024 Apr;70(2):142-148. doi: 10.1016/j.jphys.2024.02.002. Epub 2024 Mar 11. PMID 38472049
- [Derived] Theodorsen NM, Fersum KV, Moe-Nilssen R, Bo K, Haukenes I. Effect of a specific exercise programme during pregnancy on diastasis recti abdominis: study protocol for a randomised controlled trial. BMJ Open. 2022 Feb 4;12(2):e056558. doi: 10.1136/bmjopen-2021-056558. PMID 35121606